CLINICAL TRIAL: NCT06392841
Title: Hispanic/Latino and Non-Hispanic BlAck Patients Treated With niRaparib and Abiraterone Acetate Plus Prednisone for Metastatic hOrmone Sensitive Prostate Cancer With Deleterious Homologous recombinatioN Repair Alterations: a Phase II, Open Label studY
Brief Title: Niraparib, Abiraterone Acetate and Prednisone for mHSPC With Deleterious Homologous Recombination Repair Alterations
Acronym: HARMONY
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder withdrew funding.
Sponsor: Qian Qin (Other)
Collaborators: UT Southwestern Comprehensive Cancer Center (Unknown); Janssen, LP (Industry)
Responsible Party: Sponsor-Investigator, Qian Qin, Assistant Professor, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN-GU23-626
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer (mHSPC); Deleterious HRR Gene Mutation; BRCA1 Gene Mutation; BRCA2 Gene Mutation; BRIP1 Gene Mutation; CHEK2 Gene Mutation; FANCA Gene Mutation; PALB2 Gene Mutation; RAD51B Gene Mutation; RAD54L Gene Mutation
MeSH Terms: interventions — Androgen Antagonists; niraparib; Abiraterone Acetate; Prednisone; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Initial Treatment (Cycle 1 to Cycle 6) (Experimental): Androgen Deprivation Therapy (ADT) with a GnRH agonist or antagonist per standard of care. 200 mg niraparib and 1,000 mg abiraterone acetate dual action tablet (DAT, Akeega) once daily, with 5mg prednisone once daily for 24 weeks (6 cycles) unless there is progression or unacceptable toxicity. After 6 cycles, disease evaluation performed.
  Interventions: Drug: Androgen Deprivation Therapy (ADT); Drug: Niraparib/Abiraterone Acetate DAT; Drug: Prednisone
- Cohort A: prostate specific antigen (PSA) >4 ng/mL without progression at the completion of 24 weeks (Experimental): After 6 cycles, there will be an option to:
  1. Continue ADT + niraparib/abiraterone acetate plus prednisone in 28-day cycles for a total of 2 years OR until disease progression or unacceptable toxicity. Subsequent therapy will be at the discretion of the investigator per standard of care.
  2. Discontinue niraparib. Continue ADT, start abiraterone acetate plus prednisone and docetaxel 75mg/m2 in 21-day cycles. Docetaxel every 3 weeks x 6 doses. At the completion of docetaxel, the subject will move to follow-up per protocol. Niraparib should not be restarted at the completion of docetaxel. Subsequent therapy will be at the discretion of the investigator per standard of care.
  Interventions: Drug: Androgen Deprivation Therapy (ADT); Drug: Niraparib/Abiraterone Acetate DAT; Drug: Abiraterone Acetate; Drug: Prednisone; Drug: Docetaxel
- Cohort B: PSA ≤ 4 ng/mL without progression at the completion of 24 weeks (Experimental): Continue ADT + niraparib/abiraterone acetate plus prednisone for 1 year unless progression or unacceptable toxicity. At 1 year, disease evaluation will occur.
  * PSA ≥ 0.2 ng/mL: ADT + niraparib/abiraterone acetate plus prednisone will continue for 2 years or until progression or unacceptable toxicity. Therapy beyond 2 years will be per standard of care per investigator discretion.
  * PSA < 0.2 ng/mL and PSA not trending up:
    1. Continue ADT + niraparib/abiraterone acetate plus prednisone for 2 years or until progression or unacceptable toxicity. Therapy beyond 2 years will be per standard of care per investigator discretion OR
    2. STOP ADT + niraparib/abiraterone acetate plus prednisone only IF:
       * C14 PSA < 0.2 AND not trending up
       * Subjects not eligible that elect to stop ADT + niraparib/abiraterone acetate plus prednisone, will be removed from protocol treatment and move to follow-up. Subsequent therapy re-initiation will be at the discretion per standard of care.
  Interventions: Drug: Androgen Deprivation Therapy (ADT); Drug: Niraparib/Abiraterone Acetate DAT; Drug: Prednisone

INTERVENTIONS:
Drug: Androgen Deprivation Therapy (ADT) — Medical castration per ADT with GnRH agonist or antagonist (or surgical castration per orchiectomy)
Drug: Niraparib/Abiraterone Acetate DAT — Niraparib 200 mg/ Abiraterone acetate 1000 mg orally
  Other Names: Akeega
Drug: Abiraterone Acetate — 1000 mg orally
  Other Names: Zytiga
  Arms: Cohort A: prostate specific antigen (PSA) >4 ng/mL without progression at the completion of 24 weeks
Drug: Prednisone — 5 mg orally
  Other Names: Rayos; Deltasone; Prednisone Intensol
Drug: Docetaxel — 75 mg/m2 IV
  Other Names: Docefrez; Taxotere
  Arms: Cohort A: prostate specific antigen (PSA) >4 ng/mL without progression at the completion of 24 weeks

SUMMARY:
This is an open label, phase II trial in subjects with treatment naïve, metastatic hormone sensitive prostate cancer (mHSPC) with deleterious homologous recombination repair (HRR) alteration(s). These include pathologic alterations in BRCA 1/2, BRIP1, CHEK2, FANCA, PALB2, RAD51B, and/or RAD54L. A total of 64 people will be enrolled to the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. ≥ 18 years of age at the time of consent.
3. Self-identify as Hispanic/Latino or non-Hispanic black racial/ethnic background.
4. ECOG Performance Status of ≤ 2 within 30 days prior to registration.
5. Histologically confirmed diagnosis of prostate adenocarcinoma.
6. Deleterious HRR alteration(s) per any validated test, next generation sequencing (NGS) mutational analysis (tissue or liquid). These include BRCA 1/2, BRIP1, CHEK2, FANCA, PALB2, RAD51B, and/or RAD54L.
7. Radiographic evidence of metastatic disease as per conventional CT or MRI of chest, abdomen pelvis and bone scan, according to RECIST version 1.1 criteria in subjects with measurable disease and PCWG3 criteria for subjects with bone only disease (1, 2). Evidence of metastatic disease detected on Axumin or PSMA PET/CT will need confirmation on conventional CT or MRI/bone scans.
8. Hormone sensitive, treatment naïve/minimally treated [first generation androgen receptor inhibitor (ARI) such as bicalutamide ≤ 45 days, ADT ± abiraterone acetate plus prednisone ≤ 45 days allowed]. Prior therapy for localized prostate cancer allowed (including but not limited to radiation therapy, prostatectomy, lymph node dissection ± ADT, must have been completed > 6 months prior to registration).
9. Demonstrate adequate organ function as defined below. All screening labs to be obtained within 30 days prior to registration.

   * Platelets (Plt): ≥ 100 x 10^9/L (Independent of transfusions for at least 28 days prior to registration)
   * Absolute Neutrophil Count (ANC): ≥ 1.5 x 10^9/L (Independent of hematopoietic growth factors for at least 28 days prior to registration)
   * Hemoglobin (Hgb): ≥ 9 g/dL (Independent of transfusions for at least 28 days prior to registration)
   * Creatinine: Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min
   * Total bilirubin: ≤ 1.5 × ULN or direct bilirubin ≤ 1 x ULN (For subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin, and if direct bilirubin is ≤1.5 × ULN, subjects may be eligible.)
   * Aspartate aminotransferase (AST): ≤ 3 × ULN
   * Alanine aminotransferase (ALT): ≤ 3 × ULN
   * Serum potassium: ≥ 3.5 mmol/L
10. Males able to father a child who are sexually active with a female of childbearing potential must be willing to abstain from penile-vaginal intercourse or use an effective method(s) of contraception.
11. Able to swallow the study medication tablets whole.
12. Life expectancy ≥ 12 months.
13. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

1. Prostate cancer variants including predominant neuroendocrine features and/or predominant small cell carcinoma of the prostate are excluded.
2. Prior treatment with the following is excluded: second generation ARIs such as apalutamide, enzalutamide, darolutamide, or other investigational ARIs; oral ketoconazole as antineoplastic treatment for prostate cancer (allowed if total time on ketoconazole as prostate cancer-directed therapy is ≤ 10 days and discontinued prior to study treatment initiation); chemotherapy or immunotherapy for prostate cancer.
3. Radiotherapy/radiopharmaceuticals within 2 weeks of registration.
4. History of severe allergic anaphylactic reactions to niraparib/abiraterone acetate tablets or any of their excipients.
5. Current evidence of any medical condition that would make prednisone use contraindicated.
6. Long-term use of systemically administered corticosteroids (> 5mg of prednisone or the equivalent) during the study is not allowed (5mg of prednisone or equivalent daily, given with abiraterone acetate, is allowed). Short-term use of corticosteroid for indication other than in combination with abiraterone acetate (≤ 4 weeks, including taper) and locally administered steroids (eg, inhaled, topical, ophthalmic, and intra-articular) are allowed, if clinically indicated.
7. Subjects who have had major surgery ≤ 28 days prior to registration.
8. Symptomatic brain metastases.
9. Active or symptomatic viral hepatitis or chronic liver disease; encephalopathy, ascites, or bleeding disorders secondary to hepatic dysfunction.
10. Moderate or severe hepatic impairment (Class B and C per Child-Pugh classification system.
11. History of adrenal insufficiency not adequately managed.
12. History or current diagnosis of MDS/AML.
13. Current evidence within 6 months prior to registration of any of the following:

    * Severe/unstable angina, myocardial infarction, symptomatic congestive heart failure,
    * Clinically significant arterial or venous thromboembolic events (ie. pulmonary embolism), or clinically significant ventricular arrhythmias.
14. Presence of sustained uncontrolled hypertension (systolic blood pressure >160 mm Hg or diastolic blood pressure >100 mm Hg). Subjects with a history of hypertension are allowed, provided that blood pressure is controlled to within these limits by an antihypertensive treatment.
15. Human immunodeficiency virus positive subjects with 1 or more of the following:

    * Not receiving highly active antiretroviral therapy or on antiretroviral therapy for less than 4 weeks.
    * Receiving antiretroviral therapy that may interfere with the study medication
    * CD4 count <350 at screening.
    * An acquired immunodeficiency syndrome-defining opportunistic infection within 6 months of the start of screening.
    * Human immunodeficiency virus load >400 copies/mL.
16. Active infection requiring systemic therapy. NOTE: Subjects receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
17. Active malignancies (ie, progressing or requiring treatment change in the last 24 months) other than the disease being treated under study. The only allowed exceptions are:

    * Non-muscle invasive bladder cancer.
    * Skin cancer (non-melanoma or melanoma) treated within the last 24 months that is considered completely cured.
    * Malignancy that is considered cured with minimal risk of recurrence.
18. Received an investigational intervention (including investigational vaccines) or used an invasive investigational medical device within 30 days prior to C1D1.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Rate of participants with PSA decline to < 0.2 ng/ml | 24 weeks
  PSA decline is defined as percentage of participants with PSA decline to < 0.2 ng/ml at 24 weeks of therapy with ADT and niraparib/abiraterone acetate DAT plus prednisone as determined by Cycle 7 Day 1 PSA

SECONDARY OUTCOMES:
Rate of participants with PSA reduction ≥ 90% (PSA90) | 24 weeks
  Percentage of participants with PSA reduction ≥ 90% (PSA90) after 24 weeks of therapy with ADT and niraparib/abiraterone acetate DAT plus prednisone as determined by Cycle 7 Day 1 PSA
Percentage of participants with PSA decline to < 0.2 ng/ml (Cohort A) | 12 months
  Percentage of participants with PSA decline to < 0.2 ng/ml at one year in Cohort A
Percentage of participants with PSA decline to < 0.2 ng/ml (Cohort B) | 12 months
  Percentage of participants with PSA decline to < 0.2 ng/ml at one year in Cohort B (with additional evaluation of ADT + docetaxel + abiraterone acetate plus prednisone versus ADT niraparib/abiraterone acetate DAT plus prednisone)
Overall response rate (ORR) | 4 years
  Defined as the proportion of subjects achieving either a complete response or a partial response by RECIST 1.1 in subjects with measurable disease and Prostate Cancer Working Group 3 (PCWG 3) criteria for subjects with bone only metastases (1, 2)
PSA progression free survival (PFS) | 4 years
  Defined as interval from start of study treatment to the earliest event of PSA progression or death due to any cause, or the date of last known follow-up without PSA progression, whichever occurs first, according to criteria of the PCWG 3 criteria: for subjects with a decline from baseline, PSA progression is defined as the time from start of therapy to first PSA increase that is ≥ 25% and ≥ 2 ng/mL above nadir which is confirmed by a second value 3 or more weeks later (2)
Radiographic progression free survival (rPFS) | 4 years
  Defined as duration from the start of study treatment to the date of first documentation of rPFS or death due to any cause, whichever occurs first, according RECIST 1.1 in subjects with measurable disease and PCWG3 criteria for subjects with bone only disease (1, 2)
Safety of ADT and niraparib/abiraterone acetate DAT plus prednisone | 4 years
  Safety of ADT + niraparib/abiraterone acetate DAT plus prednisone through evaluation of the incidence and severity of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) as assessed by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Safety of ADT and docetaxel/abiraterone acetate plus prednisone | 4 years
  Safety of ADT + docetaxel/abiraterone acetate plus prednisone through evaluation of the incidence and severity of adverse events (AEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) as assessed by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Qian Qin, MD, Principal Investigator — UT Southwestern Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No